CLINICAL TRIAL: NCT06635018
Title: Effect of Pulse Oximeter Device on Measured Perfusion Index Values
Acronym: PICOMP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NVT_01_2024
Record Dates: First submitted 2024-10-01; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Perfusion Index
Keywords: Perfusion index; Pulse oximetry; Nociception during Anesthesia

STUDY DESIGN:
Intervention Model Description: Interventional prospective single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Determination of effect of pulse oximeters from different manufacturers on measured Perfusion index (Experimental): Three finger pulse oximeter sensors from different manufacturers are placed on the middle fingers of one hand. Three interventions subsequently follow (Resting condition, Movement artifacts and Circulation constriction).
  Interventions: Other: Resting conditions; Other: Movement artifacts; Other: Circulation constriction

INTERVENTIONS:
Other: Resting conditions — The volunteer's hands are at rest and PI readings are taken for six minutes. After two minutes, there is always a randomized rotation of the sensors between the fingers.
Other: Movement artifacts — The volunteer periodically spreads his/her fingers and clenches them into a fist, and PI readings are taken for six minutes. After two minutes there is always a randomized rotation of sensors between the fingers.
Other: Circulation constriction — The volunteer's arm is constricted using a cuff to measure non-invasive blood pressure. The perfusion index value is monitored during the time of cuff pressure and cuff release. The measurement is followed by a 4-minute pause to allow the vascular supply to stabilize, the sensors are randomly rotated, and the measurement is repeated.

SUMMARY:
The aim of this study is to experimentally determine the effect of pulse oximeters from different manufacturers on measured perfusion index values in healthy subjects at rest and with and without motion artifacts.

DETAILED DESCRIPTION:
Perfusion index (PI) is one of the many vital signs monitored to assess the clinical status of a patient. PI is determined from the pulsatile part of the plethysmographic curve, with typical values measured on the fingers ranging from 0.02% to 20%. Although PI is a relatively newly measured parameter, it has already found application in many areas of clinical medicine. It can be used as an indicator of the severity of health status in different groups of critically ill patients, e.g. in patients with sepsis, in patients after cardiac arrest, for early detection of critical heart defects, for indirect assessment of patient pain, as an indicator of fluid therapy and reactivity, or for assessment and evaluation of anaesthesia in the operating room. However, there is currently no standardised calculation of PI and different manufacturers use different algorithms for the calculation. The consequence is that absolute measured values cannot be compared between devices.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult Volunteer

Exclusion Criteria:

* Post-traumatic upper limb conditions affecting finger perfusion
* Injuries or diseases of the skin of the fingers
* Any acute phase of any disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-08 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of Perfusion Index Values Measured by Pulse Oximeters From Different Manufacturers During Rest, Movement, and Circulatory Restriction | 1 hour
  Perfusion index values will be measured and compared using pulse oximeters from different manufacturers under various conditions, including resting state, movement artifacts, and circulatory restriction. This evaluation will provide a direct comparison of the variability in perfusion index measurements across devices under each condition.

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubik, Prof., Study Chair — Czech Technical University, Fac. of Biomedical Engineering

IPD SHARING:
Plan to Share IPD: Yes
The measured data will be shared publicly in the data repository on web page: https://ventilation.fbmi.cvut.cz/data/
Supporting Information: SAP
Time Frame: Unlimited from the time of processing complete measured data
Access Criteria: Publicly available to everyone
URL: https://ventilation.fbmi.cvut.cz/data/